CLINICAL TRIAL: NCT01408316
Title: A Phase 1 Two-way Cross-over Study of the Pharmacokinetics and Pharmacodynamics of Crystalline PX-866 Tablets and Amorphous PX-866 Capsules Administered in the Fasting State, and of Crystalline PX-866 Tablets Administered Fed and Fasting, in Healthy Subjects
Brief Title: Study of the Pharmacokinetics and Pharmacodynamics of Crystalline PX-866 Tablets and Amorphous PX-866 Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PX-866-006
Record Dates: First submitted 2011-07-27; First posted 2011-08-03 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2012-03

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; PX-866; PI3K Inhibitor
MeSH Terms: interventions — PX-866

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Crystalline vs. Amorphous) (Experimental): Volunteers in part 1 of the study will initially receive either crystalline PX-866 tablets or amorphous PX-866 capsules, then after seven days, the same volunteers will respectively cross-over to receive the alternate amorphous PX-866 capsules or crystalline PX-866 tablets.
  Interventions: Drug: PX-866
- Part 2 (Crystalline Food Effect) (Experimental): Volunteers in part 2 of the study will receive two single dose treatments of PX-866 crystalline tablets initially administered in either fed or fasted state, then after at least seven days, the same volunteers will respectively cross-over to receive PX-866 tablets in the alternate fed or fasted state.
  Interventions: Drug: PX-866

INTERVENTIONS:
Drug: PX-866 — Volunteers in part 1 of the study will receive two single dose 8 mg treatments of PX-866 (one each of crystalline PX-866 tablets and amorphous PX-866 capsules) in Periods A and B, separated by at least seven days. Volunteers in part 2 of the study will receive two single dose 6 mg treatments of PX-866 (crystalline PX-866 tablets administered in either fed or fasted state), in Periods C and D, separated by at least seven days.

SUMMARY:
This is a two part study designed to evaluate the PK profile of PX-866 capsules versus tablets, and to evaluate the effect of food on the PK of PX-866 tablets only in healthy volunteers.

DETAILED DESCRIPTION:
This is a two part, Phase 1, open label, cross over study designed to evaluate the PK profile of crystalline PX-866 tablets relative to that of amorphous PX-866 capsules and to evaluate the effect of administration with food on the PK of crystalline PX-866 tablets in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age (inclusive
* Able to communicate well with study staff and to read, understand, sign and date the written informed consent form (ICF) for this study.
* Must be willing to use double barrier contraception until 90 days after last dose of study drug.
* If female and of child bearing potential, volunteer must have a negative serum pregnancy test at screening and on Day 1 or Day 1.
* Body mass index (BMI) is between 18 and 32 kg/m2 (inclusive) at screening.
* Judged by the investigator to be in good health for the purposes of this study, based on results of medical history, physical examination, ECG and laboratory testing which show no major or clinically significant findings at pre dose on Day 1.
* Has normal hepatobiliary enzyme and bilirubin (total and conjugated) results on Day 1 and/or on Day 1.
* Has normal hemoglobin, hematocrit, absolute neutrophil count, absolute lymphocyte count and platelet count on Day 1 or Day 1.
* Blood pressure is between 95 and 140 mm Hg (inclusive) systolic, 50 to 90 mm Hg (inclusive) diastolic, and pulse rate (determined by vital signs measurement) is between 40 and 100 beats per minute (inclusive) at screening and pre dose on Day 1.
* Ability and intent to comply with all requirements of the study.
* Signed ICF prior to the conduct of any study procedure.

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator, may compromise the integrity of the study data or pose a significant risk in administering study drug to the subject. This may include but is not limited to a history of relevant drug allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; or history of mental illness.
* Use of prescription medication (with systemic exposure) within 14 days prior to Day 1, or likelihood of needing to use such medication during the course of study participation.
* Use of over the counter products with systemic exposure (e.g., oral medications, herbal preparations, dietary supplements - excepting acetaminophen at less than two gm per day and vitamin supplements at or near recommended daily allowances) within 7 days prior to Day 1, or likelihood of needing to use such products during the course of study participation.
* Use of any known inhibitors or inducers of CYP3A4, (e.g., St. John's Wort, ginkgo biloba, garlic supplements, grapefruit or grapefruit juice, apple juice, or orange juice) within 7 days prior to Day 1.
* Typically consumes more than two units of alcoholic beverages per day or more than 14 units per week (one unit of alcohol being one pint [568 mL] of beer or lager, one glass [125 mL] of wine, one 25 mL shot of 40% spirits).
* Has consumed alcohol within 72 hours prior to dosing on Day 1.
* Typically consumes more than five 8 ounce servings per day of coffee, cola, or other caffeinated beverages or products with similar amounts of caffeine.
* Has consumed caffeinated beverages or products within 48 hours prior to Day 1 dosing.
* Has history of drug or alcohol abuse or addiction (by DSM IV criteria) within 2 years prior to Day 1.
* Has used tobacco or other nicotine containing product within 6 months prior to Day 1.
* Has positive urine drug screen for opiates, methadone, cannabinoids, cocaine, amphetamines/methamphetamines, barbiturates, benzodiazepines, cotinine or alcohol at the screening visit or on Day 1.
* Has participated in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 half lives (whichever is longer) prior to Day 1.
* Has been dosed with PX 866 previously.
* Has donated blood or had a significant loss of blood within 56 days prior to Day 1 or has donated more than one unit of plasma within 7 days prior to Day 1.
* Has a positive result at screening for hepatitis B antigen, hepatitis C virus antibody, human immunodeficiency virus 1 antibody or human immunodeficiency virus 2 antibody.
* Has had an illness within 5 days prior to Day 1.
* Is female and pregnant, nursing, or planning to become pregnant during the study or within 90 days of the last dose of study drug.
* Has a history of gall bladder disease, bowel pattern of ≥ 2 stools per day or intermittent diarrhea, or alteration of gastrointestinal anatomy that, in the opinion of the investigator, may alter absorption or elimination of PX 866.
* Has QTcF > 450 msec on any ECG prior to Day 1 dosing.
* In estimation of the investigator, volunteer has significant numbers of premature atrial or ventricular premature beats or other significant ECG findings, seen on continuous ECG data acquired between admission and enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax, Tmax, AUC, and T1/2 of plasma concentrations of PX-866 and PX-866 metabolites | 9 days
  Part 1: To evaluate and compare the pharmacokinetic (PK) profiles (of PX 866 and metabolites) after administration of crystalline PX 866 tablets and amorphous PX 866 capsules.
  Part 2: To evaluate the effect of food on the PK profile of crystalline PX 866 tablets.

SECONDARY OUTCOMES:
Incidence and severity of adverse events, vital signs, clinical laboratory, and ECG changes or abnormalities | 16 days
  To evaluate the safety and tolerability of crystalline PX-866 tablets.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Quint, MD, Principal Investigator — Comprehensive Clinical Development NW
Locations (1):
- Comprehensive Clinical Development NW, Tacoma, Washington, United States